CLINICAL TRIAL: NCT06813118
Title: A RCT Comparing the Effectiveness of a Combination Therapy of Lezra and Clomid Versus Lezra Alone for Inducing Ovulation in Women Diagnosed With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome
Brief Title: Comparison of Clomid and Lezra With Lezra for Ovulation Induction in Clomid Resistant PCOS Case
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rukhsana Shaheen Afzal, Assistant Professor, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HITECIMSTAXILLA
Record Dates: First submitted 2024-09-13; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene; Letrozole; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: randomization intervention RCT
Who Masked: Participant
Masking Description: lottery method for selection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental): clomiphene citrate and letrozole combination
  Interventions: Drug: Clomiphene Citrate and letrozole
- group 2 (Experimental): letrozole alone
  Interventions: Drug: Clomiphene Citrate and letrozole

INTERVENTIONS:
Drug: Clomiphene Citrate and letrozole — clomiphene citrate 100mg once daily along with letrozole 5mg to one group and letrozole 5mg to second group
  Other Names: drugs

SUMMARY:
Clomiphene citrate resistant i.e failure to ovulate after 6 cycles of ovulation induction effects 15-40% of patients with PCOS.Two treatment groups will be formed one recieving letrozole alone and another recieving CC and letrozole combined.Mature follicles and endometrial thickness will be checked by transvaginal ultrasound and results will be recorded.

DETAILED DESCRIPTION:
Subfertility is characterized by the inability to achieve conception despite engaging in regular unprotected sexual intercourse for 1-2 years.PCOS exhibits chacteristic traits such as obesity,heightened insulin resistance accompanied by compensatory hyperinsulinemia,oligo/anovulation and subfertility.Clompiphene citrate induces ovarian stimulation.Letrozole ,an aromatase inhibitor emerges as a novel medication with comparable efficacy to CC as a first line treatment for inducing ovulation in cases of anovulation.

ELIGIBILITY:
Inclusion Criteria:

* women of 20-40 years with a history of PCOS and resistant to CC

Exclusion Criteria:

* Premature ovarian insufficiency
* Husband has oligo azoospermia
* Hypothyroidism
* Hyperprolactinemia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of ovulation | 6 months
  To compare the rate of ovulation between letrozole alone and letrozole and CC

CONTACTS AND LOCATIONS:
Overall Officials: Rukhsana Shaheen Afzal, MBBS,FCPS, Principal Investigator — HITEC-Institute of Medical Sciences
Locations (1):
- HIT Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No